CLINICAL TRIAL: NCT03979625
Title: Prognosis Related to Induced Thrombopenia With Heparin Under Venoarterial ECMO in Reanimation
Acronym: TIH ECMO
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS 2016/TIH ECMO-KIMMOUN/SR
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Heparin-induced Thrombocytopenia
MeSH Terms: interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hospitalization for more than 3 days with high clinical suspicion of HIT and positive anti-PF4/heparin antibodies — Patients are classified according to results of functional tests as having either Confirmed or Excluded HIT.

SUMMARY:
Thrombocytopenia is a frequent and serious adverse event in patients treated with veno-arterial extracorporeal membrane oxygenation (VA-ECMO) for refractory cardiogenic shock. Similarly to postcardiac surgery patients, heparin-induced thrombocytopenia (HIT) could represent the causative underlying mechanism. However, the epidemiology as well as related mortality regarding HIT and VA-ECMO remains largely unknown. The investigators aimed to define the prevalence and associated 90-day mortality of HIT diagnosed under VA-ECMO.This retrospective study included patients under VA-ECMO from 20 French centers between 2012 and 2016.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient hospitalized in intensive care for a cardiovascular failure requiring the setting up of an ECMO-VA
* ECMO-VA duration ≥ 3 days
* HIT confirmed by immunological tests
* Patient affiliated to a Social Security scheme

Exclusion Criteria:

* Known antecedent of TIH prior to cannulation
* Pregnant woman
* ECMO-VA following cardiopulmonary arrest or septic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care for cardiogenic shock requiring cardiac assisting with ECMO-VA.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Death | 90 days after inclusion